CLINICAL TRIAL: NCT01196494
Title: Prospective, Controlled, Randomized Study of Intraoperative Colonic Irrigation vs. Stent Placement in Obstructive Left-Sided Colonic Cancer
Brief Title: Study of Intraoperative Colonic Irrigation Versus Stent Placement in Obstructive Left-Sided Colonic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: STENTCSPT01
Record Dates: First submitted 2010-09-07; First posted 2010-09-08 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2005-01

CONDITIONS: Colon Neoplasm; Colorectal Surgery; Intestinal Obstruction
Keywords: Obstructive left-sided colonic cancer; Colorectal stent; Intraoperative colon lavage; Lavage; Stent
MeSH Terms: conditions — Colonic Neoplasms; Intestinal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intraoperative colon lavage (Experimental)
  Interventions: Procedure: intraoperative colon lavage with primary anastomosis
- stent and deferred surgery (Active Comparator)
  Interventions: Procedure: intraoperative colon lavage with primary anastomosis

INTERVENTIONS:
Procedure: intraoperative colon lavage with primary anastomosis — Patients with obstructive left-sided colonic cancer in wich treatment in one stage procedure is intraoperative colon lavage with primary anastomosis to avoid Hartamnn´s Procedure

SUMMARY:
INTRODUCTION: There are several alternatives for one-stage emergency treatment of obstructive left-sided colonic cancer (OLCC): subtotal colectomy, intraoperative colon lavage (IOCL) with primary anastomosis, and the placement of a stent as a temporary measure prior to scheduled surgery. At present, it is not clear whether emergency perioperative lavage or the placement of a stent is the better technique. The hypothesis is that IOCL and primary anastomosis is equal safe or even safer than placement of a stent as a temporary measure prior to scheduled surgery, less length of stay and less cost.

OBJECTIVE: To establish which of these two techniques is more efficient in OLCC from the point of view of morbimortality, economic cost, and long-term survival.

MATERIAL AND METHODS:

Prospective, controlled, randomized study of patients diagnosed with OLCC. Patients were divided into two groups: group 1: stent and deferred surgery; group 2: emergency IOCL. A simple randomization system was used. The estimated sample size required per group was 21 patients. Demographic variables, risk prediction models, postoperative morbimortality, staging, complications due to the placement of stent, surgical time, clinical follow-up, health costs and follow-up of survival were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 diagnosed with complete intestinal obstruction due to tumor in the left colon using abdominal CT scan

Exclusion Criteria:

* Unresectable lesion (intraoperative), severe ischemia or cecal perforation, fecal or advanced purulent peritonitis, hemodynamic instability during surgery, immunodepressed state (corticoids, chemotherapy, HIV, major surgery in the last two months) and septic shock.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Alcantara M, Serra-Aracil X, Falco J, Mora L, Bombardo J, Navarro S. Prospective, controlled, randomized study of intraoperative colonic lavage versus stent placement in obstructive left-sided colonic cancer. World J Surg. 2011 Aug;35(8):1904-10. doi: 10.1007/s00268-011-1139-y. PMID 21559998